CLINICAL TRIAL: NCT01921959
Title: Effects of Postpartum Weight Loss Intervention on Partner and Offspring Weight
Brief Title: Fit Moms in Partners, Children, and Other Members
Status: Completed | Type: Observational
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Principal Investigator, Todd Hagobian, Assistant Professor, California Polytechnic State University-San Luis Obispo
Other Study IDs: RDK101926A
Record Dates: First submitted 2013-08-09; First posted 2013-08-14 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Partners of intervention women: Partners of women randomized to intervention
  Interventions: Behavioral: Intervention
- Partners of no intervention women: Partners of women randomized to control

INTERVENTIONS:
Behavioral: Intervention — Postpartum women are randomized to intervention or control group
  Groups: Partners of intervention women

SUMMARY:
The purpose of this ancillary study is to determine whether a behavioral weight loss intervention for postpartum mothers (5R01DK087889-02, PI Phelan; Co-I Tate) has a positive "ripple" effect on weight and health of partners and children/offspring.

DETAILED DESCRIPTION:
Lifestyle interventions targeting overweight/obese individuals can produce positive "ripple" effects on untreated overweight partners in the home. Interestingly, ripple effects on partners' weight appear most pronounced when the interventions target women. Women, and mothers in particular, remain the primary "nutritional gatekeepers" of the home. Despite widespread recognition that motherhood is a powerful motivator for behavior changes, no study to date has examined the "ripple" effects of a postpartum Internet-based lifestyle intervention that target mothers' weight. The purpose of this ancillary study is to determine whether a behavioral weight loss intervention for postpartum mothers (5R01DK087889-02, PI Phelan; Co-I Tate) has a positive "ripple" effect on weight and health of partners and children/offspring. The proposed study is ancillary to an ongoing clinic-randomized trial examining the efficacy of an innovative multicomponent (online, face-to-face, mobile phone) postpartum behavioral weight loss intervention in 408 low-income women in the Women, Infants, and Children program. The proposed study will determine whether partners of women randomized to the postpartum BWL intervention have greater weight losses and greater improvements in health outcomes than partners of women in standard WIC. Similar to the parent grant, assessments will occur at study entry, 6 months, and 12 months. This project is highly innovative, as it capitalizes on existing funded research and is the first study to examine ripple effects of multicomponent Internet-based intervention in low-income individuals. The project also has high impact, as the postpartum period is a powerful motivator for behavior and environmental changes in the home; and, if positive ripple effects occur, the field of obesity treatment and prevention could move beyond focus on individual level to the often, unrecognized interpersonal effects of lifestyle interventions. PUBLIC HEALTH RELEVANCE: This research project will examine whether a postpartum weight-loss intervention has a positive "ripple" effects on weight and health of untreated partners and offspring/children in the home.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman who self-identifies as sharing an intimate relationship and cohabitating in the home with the postpartum woman (enrolled in the parent grant) for the previous 3 months or recently been married and living in the home
* ≥18 years
* willing to provide informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Partners of postpartum women
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Weight and Weight Change | 12 months
  Absolute weight and change in weight

CONTACTS AND LOCATIONS:
Overall Officials: Todd Hagobian, PhD, Principal Investigator — Cal Poly San Luis Obispo
Locations (1):
- California Polytechnic State University, San Luis Obispo, California, United States